CLINICAL TRIAL: NCT07201493
Title: Evaluation of New Color Temperature Adjustment Mode in Preventing Dry Eye and Visual Fatigue
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TREC2025-KY185
Record Dates: First submitted 2025-09-20; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Visual Fatigue; Dry Eye
Keywords: visual fatigue; tear break-up time; dry eye; VDT syndrome; critical flicker fusion frequency
MeSH Terms: conditions — Asthenopia; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This study is designed with a total of three groups, where participants will sequentially and randomly undergo all the intervention procedures.
Who Masked: Participant
Masking Description: In order to eliminate the influence of subjective factors during the examination, this study was blinded only to the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6500K group (No Intervention): This is the group that performs visual evoked tasks using conventional color temperature mode of whose vaule is 6500K. In this group, the impact of the same text content on the visual fatigue and comphrehensive analysis of tear film were assessed, including but not limited to indicators such as blinking detection, visual function and so on.
- sigmoid change group (Experimental): This is the group that performs visual evoked tasks using dynamic color temperature change mode 1 which changes from 6500K to 4000K. In this group, the impact of the same text content on the visual fatigue and comphrehensive analysis of tear film were assessed, including but not limited to indicators such as blinking detection, visual function and so on.
  Interventions: Behavioral: color temperature change mode
- gradient change group (Experimental): This is the group that performs visual evoked tasks using dynamic color temperature change mode 2 which changes from 6500K to 4000K. In this group, the impact of the same text content on the visual fatigue and comphrehensive analysis of tear film were assessed, including but not limited to indicators such as blinking detection, visual function and so on.
  Interventions: Behavioral: color temperature change mode

INTERVENTIONS:
Behavioral: color temperature change mode — Subjects are asked to read a terminal display device for 50 minutes, featuring texts with different color temperature mode treatments. Specifically, they will read the same text content for 50 minutes with different color temperature mode. The participants will complete a total of 2 sets of tests in a random order.
  Arms: gradient change group; sigmoid change group

SUMMARY:
The purpose of this study was to investigate the effects of visual fatigue and dry eye level under different correlated color temperature modes, and to evaluate the effect of new designed dynamic color temperature change modes on the improvement of visual fatigue and dry eye level.

DETAILED DESCRIPTION:
The effect of electronic display devices on visual fatigue of human eyes was the primary evaluation index and the primary outcome index of this experiment. Secondary outcome indicators were tear film break-up time, tear lipid analysis, conjunctival congestion score and subjective visual fatigue score. Other outcome indicators were eyeblink detection, accommodative function and Schirmer test. Baseline values of the above metrics were measured separately before each group of trials and then, after 50 minutes of e-text reading, specific values of the different metrics were collected when using different color temperature modes and all valid measurements were statistically compared and analysed. To assess the effect of new designed dynamic color temperature change modes on reducing visual fatigue and dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult population, regardless of gender.

  * Refractive error is less than or equal to -1.5D and both eyes achievecorrected visual acuity of 0.8 or higher.
  * Normal intraocular pressure with no organic pathology.
  * No apparent symptoms of dry eye.
  * Willing to cooperate to complete all the tests.
  * Voluntarily signing the informed consent form.

Exclusion Criteria:

* Individuals with strabismus and amblyopia exist.

  * Suffering from congenital eye conditions such as congenital cataracts or congenital retinal diseases.
  * Those who have undergone intraocular surgery (such as cataract removal, intraocular lens implantation, etc.).
  * Individuals with refractive media opacity (such as corneal lesions, lens opacity, etc.).
  * Only one eye meets the inclusion criteria.
  * Active corneal infections such as bacterial, fungal, viral, or other acute or chronic anterior segment inflammations.
  * Currently using medications that may lead to dry eye or affect vision and corneal curvature.
  * Other ocular conditions, such as dacryocystitis, eyelid disorders and abnormalities, abnormal intraocular pressure, and glaucoma.
  * Unable to undergo regular eye examinations.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Critical flicker fusion frequency | Participants underwent three randomized experimental conditions through study completion, an average of 1 months. For each condition, CFF test was administered at baseline (pre-experiment) and post-task,totaling six completions per participant.
  Critical flicker fusion frequency was measured before and after the task by a flicker fusion frequency detection device to assess changes in the degree of ocular fatigue. To compare the difference in CFF after wearing anti-blue glasses with normal glasses and to evaluate the effect of anti-blue glasses in preventing asthenopia.

SECONDARY OUTCOMES:
Visual fatigue | Participants underwent three randomized experimental conditions through study completion, an average of 1 months. For each condition, visual fatigue test was administered at baseline and post-task,totaling six completions per participant.
  The visual fatigue questionnaire utilized in this study consists of a self-report survey with a total of 16 items. It is designed to comprehensively assess the severity of visual fatigue symptoms, with a scoring system ranging from 0 to 4. Higher scores indicate more severe symptoms, encompassing three primary domains: ocular symptoms, visual discomfort, and psychological aspects triggered by visual fatigue.
tear break-up time | Participants underwent three randomized experimental conditions through study completion, an average of 1 months. For each condition, CFF test was administered at baseline (pre-experiment) and post-task,totaling six completions per participant.
  This clinical study included tear film breakup time measurement using keratograph-7000,OCULUS immediately after each VDT task, reflecting tear film stability, and evaluating the degree of dry eye
Measurement of Accommodative Sensitivity with Flip-Chart Post-VDT Tasks | Participants underwent three randomized experimental conditions through study completion, an average of 1 months. For each condition, CFF test was administered at baseline (pre-experiment) and post-task,totaling six completions per participant.
  This clinical study involves the assessment of accommodative sensitivity for both monocular and binocular vision using a flip-chart immediately following each VDT task. The measurement will quantify the number of optotypes correctly identified within one minute, indicative of the subject's accommodative capacity.

OTHER OUTCOMES:
equivalent refraction | Participants underwent three randomized experimental conditions through study completion, an average of 1 months. For each condition, CFF test was administered at baseline (pre-experiment) and post-task,totaling six completions per participant.
  This clinical study included testing subjects for equivalent refraction diopters, which can indirectly reflect changes in the degree of myopia in the eye after the use of VDT at close range.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University,, Beijing, Beijing/China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No